CLINICAL TRIAL: NCT07325695
Title: The Effect of Virtual Reality Glasses on Perceived Pain and State Anxiety Levels During Intrauterine Device Insertion: a Randomized Controlled Study
Brief Title: Effect of Virtual Reality Glasses on Pain and Anxiety During Intrauterine Device Insertion in Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Serap Ozturk Altinayak (Other)
Responsible Party: Sponsor-Investigator, Serap Ozturk Altinayak, Associate Professor, Ondokuz Mayıs University
Organization: Ondokuz Mayıs University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Ondokuz Mayıs Üniversitesi
Record Dates: First submitted 2025-12-09; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Pain; Anxiety
Keywords: virtual reality; anxiety; pain management
MeSH Terms: conditions — Pain; Anxiety Disorders; Agnosia

STUDY DESIGN:
Intervention Model Description: Two parallel groups wiil be compared: VR distraction during IUD insertion versus standard care control
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality Group (Experimental): Participants will wear a VR headset during IUD insertion for pain and anxiety distraction
  Interventions: Device: Virtual Reality Headset
- Control Group (No Intervention): Participants will receive standard care during IUD insertion without VR intervention

INTERVENTIONS:
Device: Virtual Reality Headset — A VR headset will be used to provide immersive distraction during intrauterine device insertion to reduce pain and anxiety
  Arms: Virtual Reality Group

SUMMARY:
This study aims to evaluate the effect of virtual reality glasses on pain perception and anxiety levels during intrauterine device insertion in women. Participants undergoing intrauterine device insertion will be randomly assigned to either a virtual reality invervention group or a standard care control group. Pain intensity and anxiety levels will be assessed during and after the procedure using validated measurement tools. The findings of this study may contribute to improving patient comfort during intrauterine device insertion.

DETAILED DESCRIPTION:
This randomized controlled study will be conducted among women scheduled for intrauterine device insertion. Eligible participants will be randomly allocated into two groups: a virtual reality intervention group and a control group receiving standard care. Participants in the intervention group will be use virtual reality glasses during the intrauterine device insertion procedure, while the control group will undergo the procedure without virtual reality. Pain intensity will be measured using a validated pain scale during and after the procedure. Anxiety levels will be assessed using a validated state anxiety measurement tool. Sociodemographic and clinical characteristics of participants will also be recorded. The study will be conducted in accordance with ethical principles, and informed consent will be obtained from all participants.

ELIGIBILITY:
Inclusion Criteria:

* Those aged 18-49
* Those who understand and speak Turkish
* Those without visual or hearing impairments
* Women who agree to participate in the study
* Those with adequate mental and emotional health
* Those who will undergo a copper intrauterine device (IUD)

Exclusion Criteria:

* Those outside the 18-49 age range
* Those who do not speak Turkish
* Those with visual, hearing, or speech impairments
* Those with diagnosed psychiatric illnesses
* Those taking psychiatric medications

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — This study is based on a female-specific reproductive health intervention(İntrauterine device placement
Enrollment: 70 (Actual)
Dates: Start 2025-03-04 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
Pain insensity during IUD insertion | İmmediately after the procedure
  Pain severity will be measured immediately after the IUD insertion procedure using the Visual Analog Scale
Pain catastrophizing(Pain Catastrophizing Scale, PCS) | İmmediately after the procedure
  Pain catastrophizing will be assessed immediatel the IUD insertion procedure using the Pain Catastrophizing Scale(PCS;13 items). Higher scores indicate greater catastrophizing.
State Anxiety level(STAI-S) | İmmediately after the procedure
  State anxiety will be measured immediately after the procedure using the State-Trait Anxiety Inventory- State Subscale(STAI-S). Higher scores indicate greater anxiety.

CONTACTS AND LOCATIONS:
Locations (1):
- Ondokuz Mayis University, Samsun, Samsun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
No individual participant data will be shared